CLINICAL TRIAL: NCT01819454
Title: The Diagnostics of Extraesophageal Reflux With the Restech System in Patients With Chronic Rhinosinusitis
Brief Title: The Diagnostics of Extraesophageal Reflux With the Restech System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-EER Restech; NT13500-4/2012 (Other Grant/Funding Number: Internal Grant Agency Ministry of Health)
Record Dates: First submitted 2013-03-22; First posted 2013-03-27 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Nasal Diseases; Nasal Polyps; Laryngopharyngeal Reflux
Keywords: chronic rhinosinusitis; extraesophageal reflux; Restech system; antireflux therapy
MeSH Terms: conditions — Nose Diseases; Nasal Polyps; Laryngopharyngeal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- pH monitoring sinusitis no polyps (Experimental): 30 patients with chronic rhinosinusitis without nasal polyposis, without asthma bronchiale or ASA syndrome
  Interventions: Device: pH monitoring (Restech)
- pH monitoring sinusitis with polyp (Experimental): 30 patients with chronic rhinosinusitis with nasal polyposis, without asthma bronchiale or ASA syndrome
  Interventions: Device: pH monitoring (Restech)
- pH monitoring sinusitis, polyps, asthma (Experimental): 30 patients with chronic rhinosinusitis with nasal polyposis and with asthma bronchiale and/or ASA syndrome
  Interventions: Device: pH monitoring (Restech)

INTERVENTIONS:
Device: pH monitoring (Restech) — see in "detail description of the study" part of the protocol
  Other Names: oropharyngeal pH monitoring using Restech system

SUMMARY:
The aim of the project is to define the frequency with which EER is present in patient with chronic rhinosinusitis (CHR). The measurement will be carried out with a 24-hour monitoring of the pH using the Restech system. This modern device is equipped with a narrow antimony probe. The sensor is able to record not only liquid but also aerosol reflux episodes. The second aim is to determine the relation among EER, CHR and asthma bronchiale. We will compare the presence of reflux in three different patient groups (1. CHR without nasal polyposis, without asthma bronchiale or ASA syndrome, 2. CHR with nasal polyposis, without asthma bronchiale or ASA syndrome, 3. CHR with nasal polyposis and asthma bronchiale and/or ASA syndrome). We expect to find a significantly more frequent presence of EER in patients with CHR and asthma bronchiale or ASA syndrome. In case our hypothesis is confirmed, it will be especially these patients(with a difficult to manage nasal polyposis) benefiting from the antireflux therapy.

DETAILED DESCRIPTION:
Introduction The problems of relation between some of the ENT diseases (posterior laryngitis, granulomas of the vocal cords, globus pharyngeus and others) and the extraesophageal reflux (EER), which is associated by the refluxate penetrating above the level of the upper oesophageal sphincter, has been studied more intensely especially during the last several years. The golden standard in the diagnostics of EER remains the dual-channel 24-hour pH-metry. The methodology of this procedure has been standardized in the past several years and differs significantly from the oesophageal pH-metry carried out by gastroenterologists (the upper probe is usually placed above the level of the upper oesophageal sphincter). The pH-metry enables us to monitor especially the impact of EER upon diseases of the oesophagus and hypopharynx. Non-existence of a simple and sensitive method was a barrier in a more detailed examination of the relations between EER and the more proximally located parts of the upper respiratory tract (nasopharynx, nasal cavity and paranasal sinuses, middle-ear cavity). The problem of "classical" pH-metry probes lies in the fact that unless the sensor is covered by a mucosa, it dries out and the record is not accurate.

The Restech system was introduced two years ago, with the aim to improve the EER diagnostics in oropharynx and nasopharynx. The sensor of a very sensitive antimony probe is positioned at the tip of a 1,5 mm catheter, which is inserted through the nose behind the uvula (the exact positioning is controlled with the use of the illuminating end of the catheter). High sensitivity of this device enables to measure not only the pH of the liquid but also of small aerosol drops - so called aerosol reflux. The examination takes 24 hours, the data are being transferred wirelessly into a recording device. Normative data of a non-symptomatic group have also been defined. The advantages of this method, when compared with the dual-probe 24-hour pH-metry are a higher sensitivity, easier accomplishment and better compliance of the patient population. However, a wider comparison data for different pathological conditions are still missing.

EER is considered to be one of possible factors which may contribute to the onset or worsen existing chronic rhinosinusitis (CHR). It is a well-known fact that a part of the patients with CHR undergoing endonasal surgery suffer from an early recurrence of the disease. DelGaudio found out, using a 3-channel pH-metry, that adult patients with refractory or recurrent chronic rhinosinusitis experience a significantly higher number of nasopharyngeal refluxes, when compared to the patient population presenting no symptoms after surgical treatment; and recommends anti-reflux therapy as a part of treatment in patients with refractory chronic rhinosinusitis. The same view is supported by another author, Pincus, who in his clinical trial confirmed a good effect of proton pump inhibitors in the treatment of such patients. According to EPOS (European Position Paper On Rhinosinusitis and Nasal Polyps, 2007), the relation between EER and chronic rhinosinusitis is currently at the level of a III degree evidence. EPOS also summarises the fact that patients suffering from chronic rhinosinusitis and pH-metry proven EER, present significantly more frequently alleviation of the symptoms following an anti-reflux therapy. In that respect, EPOS recommends further clinical investigation of this problem.

It is possible to assume that the Restech system enables a more precise diagnostics of the patients (when compared to pH-metry), however this system has not been tested in the diagnostics of EER in patients with CHR, either in the Czech Republic or abroad. If the proposed relation is confirmed, it will mean a dramatic change in the process of treatment in a part of the CHR patients, suffering at the same time from EER ("more urgent" recommendation of anti-reflux therapy, especially in patients with recurrent and refractory CHR).

It has been proved in the past that a part of the patient population with difficult to control asthma bronchiale also suffers from EER, and that these patients profit greatly from a treatment using proton pump inhibitors. Also a part of the patients with CHR suffers from asthma bronchiale or a complete ASA syndrome. It is possible to assume that EER, having a negative impact upon the asthma bronchiale, may have a similar negative effect upon CHR. The mutual interrelations among EER, CHR and asthma bronchiale have not been thoroughly studied; one of the aims of the proposed project is also to explore these relations.

Aims of the project

* to determine how often is EER present in the patient population with CHR
* to compare the occurrence of EER in three groups of patients

  1. CHR without nasal polyposis, without asthma bronchiale or ASA syndrome
  2. CHR with nasal polyposis, without asthma bronchiale or ASA syndrome
  3. CHR with nasal polyposis and asthma bronchiale and/or ASA syndrome

Working hypotheses

1. A part of the patients with CHR present with a significant pathological EER penetrating into nasopharynx (significantly higher number of EER episodes, when compared with asymptomatic population)
2. EER is more frequent in patients with CHR and concomitant asthma bronchiale or ASA syndrome

Methodology The project is designed as a prospective study which is in compliance with the principles and policies of the Helsinki Declaration and has been approved by the Ethics Committee.

Patients: The patients will be enrolled into the study at the rhinology out-patient part of the ENT department of the University Hospital Ostrava.

A total of 90 patients will be enrolled into the study within 4 years: 30 patients suffering from CHR without nasal polyposis, without asthma bronchiale or ASA syndrome, 30 patients suffering from CHR with nasal polyposis, without asthma bronchiale or ASA syndrome, and 30 patients suffering from CHR with nasal polyposis and asthma bronchiale and/or ASA syndrome Inclusion criteria: 1/ age (18-60 years), 2/ signing of the informed consent. Entry examination: Patients enrolled into the study will be asked to complete a questionnaire (age, sex, body weight, body height, smoking habits, asthma bronchiale or ASA syndrome, the period of treatment for CHR, the number of endonasal surgeries in the past), and further will complete the Reflux symptom questionnaire (questionnaire used to determine the symptoms typical for EER), Reflux finding score (findings in the larynx typical for EER) and the degree of polyposis (1.-3.) will be recorded.

24-hour monitoring of the nasopharyngeal pH using the Restech system: Description of the Restech device please see "Introduction". The measure parameters to prove EER in the nasopharyngeal area: the number of EER episodes, fractional time below pH 5.5 and RYAN composite score.

Data collection, analysis of data and proposal of the statistical processing The statistical processing will be carried out by Ing. Hana Tomášková, PhD. from the Institute of Epidemiology and Public Health, Medical Faculty of the Ostrava University.

1. The percentage of patients with EER will be defined from the overall number of CHR patients and individually for each group.
2. We will determine whether there exists a significantly higher percentage of patients with EER in any of the three examined groups, when compared with the other groups.
3. Other independently assessed factors in the group of patients with proven EER and the group without proven EER will be the age, sex, BMI, smoking habits, Reflux symptom index, Reflux finding score, asthma bronchiale or ASA syndrome, the length of CHR treatment, the number of endonasal surgeries in the past and the degree of nasal polyposis.

The method of descriptive statistics will be used for statistical processing (arithmetic mean, standard deviation, frequency tables), X2 test, Fisher's exact test, analysis of variance (ANOVA), OR calculation (odds ratio) with 95% confidence intervals and logistic regression. The statistical tests will be assessed on the significance level of 5%. The statistical analysis will be carried out with the Stata v. 10 programme. We will use the MS Excel programme for data collection.

Discussion Measurement of pH with the Restech system is a new and sophisticated method which has been introduced into the clinical practice in the course of the past two years. The first normative data and composite RYAN score have already been defined for healthy population (please see Literature). Now it is necessary to verify the correlations with symptoms and clinical findings in different patient groups, which may be worsened by EER. One of such patient groups are also patients with CHR. There are just a few sparse publications in the world literature (DelGaudio, Pincus) examining the relation between EER and CHR with the use of pH-metry. These studies suggest the fact that EER may be considered a negative prognostic factor from the point of view of an early recurrence of nasal polyposis after an endonasal surgery. Also EPOS recommends further studies to be conducted regarding this topic. The aim of the proposed work is to define, using the measurement of nasopharyngeal pH with the Restech system (which is more accurate and sensitive than pH-metry), how often is a pathological EER present in patients with CHR. At the same time we will determine the relation among EER, CHR and asthma bronchiale. A clinical trial such as this does not exist in the world literature so far. In case we confirm the relation between CHR and EER, the clinical impact will be significant, taking into consideration the number of patients with CHR.

Benefits of the project In case we confirm the hypothesis that EER is significantly more present in patients with CHR when compared to the common population, it is possible to expect that the antireflux therapy may be introduced into the treatment protocol of these patients. The presumption is such that the anti-reflux treatment will alleviate the patients´ symptoms (nasal patency, secretion), and possibly also decrease the number of recurrences and necessary reoperations. This will decrease the risks related to surgical procedures and improve the quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* signing of the informed consent
* patients with chronic rhinosinusitis

Exclusion Criteria:

-non-tolerance of the pH catheter

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-08; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The frequency of the extraesophageal reflux in patients with chronic rhinosisnusitis | 3 years
  EER will be measured using RYAN score, number of episodes and time of pH below 5.5

CONTACTS AND LOCATIONS:
Overall Officials: Karol Zelenik, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

REFERENCES:
- [Background] DelGaudio JM. Direct nasopharyngeal reflux of gastric acid is a contributing factor in refractory chronic rhinosinusitis. Laryngoscope. 2005 Jun;115(6):946-57. doi: 10.1097/01.MLG.0000163751.00885.63. PMID 15933499
- [Background] Katle EJ, Hatlebakk JG, Steinsvag S. Gastroesophageal reflux and rhinosinusitis. Curr Allergy Asthma Rep. 2013 Apr;13(2):218-23. doi: 10.1007/s11882-013-0340-5. PMID 23371037
- [Background] Loehrl TA, Samuels TL, Poetker DM, Toohill RJ, Blumin JH, Johnston N. The role of extraesophageal reflux in medically and surgically refractory rhinosinusitis. Laryngoscope. 2012 Jul;122(7):1425-30. doi: 10.1002/lary.23283. Epub 2012 Apr 26. PMID 22539181
- [Background] Hanna BC, Wormald PJ. Gastroesophageal reflux and chronic rhinosinusitis. Curr Opin Otolaryngol Head Neck Surg. 2012 Feb;20(1):15-8. doi: 10.1097/MOO.0b013e32834e8f11. PMID 22157165
- [Derived] Zelenik K, Matousek P, Formanek M, Urban O, Kominek P. Patients with chronic rhinosinusitis and simultaneous bronchial asthma suffer from significant extraesophageal reflux. Int Forum Allergy Rhinol. 2015 Oct;5(10):944-9. doi: 10.1002/alr.21560. Epub 2015 Jun 5. PMID 26046448